CLINICAL TRIAL: NCT01738997
Title: Endoscopical Dilation of Benign Esophageal Strictures - a Randomized, Clinical Trial, Comparing Two Different Inflation Times.
Brief Title: Endoscopical Dilation of Benign Esophageal Strictures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Umeå (Other)
Collaborators: Uppsala University (Other); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Bengt Wallner, MD, PhD, University Hospital, Umeå
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 02-499
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Dysphagia
Keywords: Benign; Esophageal strictures; Esophagus; Balloon Dilation
MeSH Terms: conditions — Deglutition Disorders; Esophageal Stenosis | interventions — Dilatation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Dilation 10 sec
  Interventions: Device: Dilation 10 sec
- Group B (Active Comparator): Dilation 2 min
  Interventions: Device: Dilation 2 min

INTERVENTIONS:
Device: Dilation 10 sec
  Other Names: CRE, Controlled Radial Expansion, Boston Scientific Cork Ltd
  Arms: Group A
Device: Dilation 2 min
  Other Names: CRE, Controlled Radial Expansion, Boston Scientific Cork Ltd
  Arms: Group B

SUMMARY:
Although balloon dilatation is the primary treatment for benign dysphagia, information about the optimal inflation time is lacking. The aim of the current pilot study was to compare 10 seconds inflation time, with 2 minutes inflation time, regarding the efficacy

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic dysphagia with an endoscopic picture suggestive of a benign disease

Exclusion Criteria:

* Suspicion of achalasia or malignancy. If the patients needed more than 3 dilations the first month this was also a considered an exclusion criterion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-12; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Relief from dysphagia | 1 year from dilation